CLINICAL TRIAL: NCT00929942
Title: Treatment of Benign Bronchial Airway Stenoses in Patients After Lung Transplantation With a Biodegradable Stent - a Proof of Concept Study
Brief Title: Biodegradable Stents in Lung Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: ELLA-CS, Czech Republic (Unknown)
Responsible Party: Karel Volenec, ELLA-CS, s.r.o.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5237
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2009-06

CONDITIONS: Lung Transplantation
Keywords: lung transplantation; bronchial stenosis; biodegradable stent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DV Stent (Experimental): Intervention "SX-ELLA Stent Degradable DV Bronchial (DV Stent)" will be implanted in the target lesion in general anesthesia under fluoroscopy or by direct vision. Before dilatation, extension of the airway complications will be measured by bronchoscopy and documented.
  Interventions: Device: SX-ELLA Stent Degradable DV Bronchial (DV Stent)

INTERVENTIONS:
Device: SX-ELLA Stent Degradable DV Bronchial (DV Stent) — Intervention "SX-ELLA Stent Degradable DV Bronchial (DV Stent)" will be implanted in the target lesion in general anesthesia under fluoroscopy or by direct vision. Before dilatation, extension of the airway complications will be measured by bronchoscopy and documented.

SUMMARY:
A prospective observational trial involving 10 patients is planned. Intervention "SX-ELLA Stent Degradable DV Bronchial (DV Stent)" will be implanted in the target lesion in general anesthesia under fluoroscopy or by direct vision. Before dilatation, extension of the airway complications will be measured by bronchoscopy and documented.

DETAILED DESCRIPTION:
Obstructive airway complications (OAC) (bronchial stenosis) are a significant problem in lung transplantation (LTx), and a special subset of chronic graft dysfunction. The overall rate is approximately 20% per recipient. Even though disobliteration (laser, argon-coagulation, cryotherapy) or balloon dilatation (bronchoplasty) are performed there is a high rate of recurrence. Self expandable metallic stents (SEMS) is one suggested treatment option after failed initial therapy but have a high rate of re-stenosis (50-60%). Morbidity, the risk for e.g. infection and atelectasis and lower long-term survival are often consequences in pts. treated with SEMS. No surgical options aside from re-do-transplantation are available. OAC are developing mostly in the time 3 - 6 months post Tx. The idea is a permanent but temporary therapy with replacement character of the stenosis which is given in degradable bronchial stents.

Hypothesis: New biodegradable bronchial stents are a successful treatment of benign bronchial stenosis after lung transplantation. After stent placement is further disobliteration is less frequently used during the next 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent airway complication (obstructive or necrotic) after single-order double-lung transplantation (at least twice balloon-dilatation or disobliteration therapy).
* Patient at least 3 months after lung transplantation and followed in MHH outpatient clinic.
* Target lesion in the left or right main stem bronchus, intermediate bronchus, right or left lower lobe, left upper lobe. Multiple lesions are eligible for inclusion and treatment but DV-stent implantation in different target lesions should be at least 6 weeks apart.

Exclusion Criteria:

* Pregnant or breast feeding women.
* Patients who are using no double-barrier method of birth control.
* Previous use of a metallic stent (SEMS).
* Target lesion in the middle lobe bronchus, right upper lobe, carina or trachea.
* Previous use of brachytherapy or topical mitomycin.
* Pats. after heart-lung transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Show that DV stent can be safely placed in LTx recipients and are effective in relief of symptoms associated with OAC. | 6 months

SECONDARY OUTCOMES:
To demonstrate mucosal healing in the first 6 months after stent insertion. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jens T Gottlieb, M.D., Principal Investigator — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany